CLINICAL TRIAL: NCT03216005
Title: Investigation of Femoropopliteal In Situ Valve Formation With the InterVene System
Acronym: INFINITE-OUS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Intervene, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLN 003
Record Dates: First submitted 2017-07-07; First posted 2017-07-12 (Actual); Last update posted 2021-09-10 (Actual); Status verified 2021-09

CONDITIONS: Chronic Venous Insufficiency

STUDY DESIGN:
Intervention Model Description: prospective, non-randomized, multicenter pre-market feasibility study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (1):
- BlueLeaf System (Experimental): The BlueLeaf System will be used to create an autogenous leaflet to mimic valve function.
  Interventions: Device: BlueLeaf System

INTERVENTIONS:
Device: BlueLeaf System — The BlueLeaf System will be used to create an autogenous leaflet to mimic valve function.

SUMMARY:
To evaluate the safety and effectiveness of the BlueLeaf System for the restoration of venous competence for the treatment of symptomatic chronic venous insufficiency (CVI).

DETAILED DESCRIPTION:
Prospective, non-randomized, multicenter pre-market feasibility study to evaluate subjects treated with the BlueLeaf System for the treatment of symptomatic CVI of the lower extremity. The BlueLeaf System is designed to form autogenous tissue leaflets from vein walls in the femoral and popliteal veins without the use of a permanent vascular implant for the treatment of CVI. Subjects meeting eligibility criteria will be enrolled and may be followed through 5 years post treatment.

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic CVI subjects, Clinical Etiological Anatomical Pathophysiological (CEAP) grade 3 to 6;
* Failed compression therapy of at least 6 months' duration;
* Deep system venous reflux characterized by >1 second reflux time;
* Presence of at least one target site within the target vessel.

Exclusion Criteria:

* Untreated significant superficial venous incompetence which, in the opinion of the Investigator, may be the primary source of existing symptoms;
* Deep venous intervention in the target limb or outflow vessels within 6 months of consent;
* Significant peripheral arterial disease with an ankle-brachial index of <0.50 or with incompressible vessels;
* Acute deep venous thrombosis (DVT) within 3 months of consent;
* History of stroke within the last 6 months;
* Flow-limiting venous outflow obstruction central to the intended target sites;
* Insufficient inflow through the treatment vein upon manual augmentation;
* Chronic, diffuse, post-thrombotic femoropopliteal vein disease that, in the Investigator's opinion, would preclude venous valve formation or would inhibit flow through the treatment sites;
* Chronic renal insufficiency with creatinine level of ≥2mg/dL;
* Hemoglobin level <9.0 mg/dL;
* Platelet count <50,000 or >1,000,000 per mm3;
* Total white blood cell count <3,000/mm3;
* Pregnant or lactating female; positive pregnancy test, women of childbearing potential must be tested;
* Non-ambulatory patients;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2017-11-02 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Percent decrease in reflux time (RT) in the primary treated vein segment from pre-procedure baseline to the 30-day follow-up imaging study | 30 days
Freedom from target vessel deep venous thrombosis (DVT) at the 30-day follow-up imaging study. | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Fletcher Wilson, Study Director — Intervene, Inc.
Locations (5):
- Australia (2):
  - Royal Prince Alfred, Camperdown, New South Wales
  - Prince of Wales, Randwick, New South Wales
- Vancouver Coastal Health Research Institute, Vancouver, British Columbia, Canada
- New Zealand (2):
  - Auckland City Hospital, Auckland
  - Clinical Trials New Zealand Ltd, Hamilton

IPD SHARING:
Plan to Share IPD: No